CLINICAL TRIAL: NCT02884141
Title: Assessment of Renal and Cervical Artery DysplasIA
Brief Title: Cross-sectional Study of Patients With Renal or Craniocervical Fibromuscular Dysplasia
Acronym: ARCADIA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de Recherche sur l'Hypertension Artérielle (Other)
Responsible Party: Sponsor
Other Study IDs: P071241-Arcadia; 2009-A00288-49 (Registry Identifier: ID-RCB (France: Agence Nationale de Securite du Medicament))
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-05

CONDITIONS: Fibromuscular Dysplasia
Keywords: Renal Artery Obstruction; Carotid Artery Diseases; Genetic Association Studies
MeSH Terms: conditions — Fibromuscular Dysplasia; Renal Artery Obstruction; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with documented fibromuscular dysplasia (see inclusion criteria).
  Non-usual care added acts:
  * blood sampling
  * urine sampling
  * renal echography

SUMMARY:
ARCADIA is a national registry designed to document phenotypic and genetic traits in patients with renal and/or cervical artery fibromuscular dysplasia (FMD).

FMD is a group of arterial diseases that most commonly involve renal and carotid arteries. Patients with FMD may present with renovascular hypertension and/or with cerebrovascular symptoms. Angiographic classification includes the multifocal type and the focal type. FMD may affect one or more vascular beds and progress to more severe stenosis and to renal or cerebrovascular complications. FMD may be familial (OMIM #135580).

Our main objective is to create a FMD registry that will collect standardized information from all consenting patients diagnosed with the condition in 16 participating centers. This registry, along with a collection of leukocyte DNA, will constitute a resource for further clinical research on FMD. The first application will be the assessment of the frequency of multi-site FMD, i.e. the frequency of cervical artery FMD in patients presenting with renal artery FMD and vice-versa. The second application will be a case-control study to identify susceptibility genes for FMD.

Patients are eligible in the registry if: (a) they have renal or cervical artery FMD with either multifocal or focal lesions at CT-angiography, MR-angiography, or intra-arterial angiography; (b) they give informed consent to leukocyte DNA analysis and to the collection of bioclinical and morphologic information. Phenotypic assessment will be performed in accordance with current recommendations and best clinical practice.

Given the multicenter nature of the study and the recruitment capacity of each centre, enrollment of 500 FMD cases is expected over 5 years. This number will 1) allow an accurate estimation of the frequency of multi-site FMD: when the sample size is 500, a two-sided 95% confidence interval will extend 0.035 from the observed proportion for an expected proportion of 0.20 based on a previous report and from our unpublished data. 2) In addition to a collection of 400 renal FMD already collected at HEGP, give sufficient power for a genome-wide association study seeking for susceptibility genes

DETAILED DESCRIPTION:
1. Background

   1. Definition

      FMD is a group of nonatherosclerotic, noninflammatory arterial diseases that most commonly involve the renal, cervical (carotid, and vertebral) arteries. Histological classification discriminates three main subtypes, intimal, medial and perimedial, which may be associated in a single patient. Angiographic classification includes the multifocal type, with multiple stenoses and the 'string-of-beads' appearance that is related to medial FMD, and tubular and focal types, which are not clearly related to specific histological lesions (unclassified FMD).

      Aneurysms and dissections are considered to be complications of FMD but frequently arise in individuals with no FMD. Therefore, their presence without direct evidence of FMD does not suffice to diagnose the condition.
   2. Presentations

      The prevalence of symptomatic renal artery FMD is about 4/1000 and the prevalence of cervical FMD is probably half that.

      Renovascular hypertension is the most common manifestation of renal artery FMD. Multifocal stenoses with the 'string-of-beads' appearance are observed at angiography in more than 80% of cases, mostly in women aged between 30 and 50 years; they generally involve the middle and distal two-thirds of the main renal artery and in some case also renal artery branches. Spontaneous renal artery dissections are rare but frequently coexist with FMD.

      Cervical FMD can be complicated by dissection with headache, Horner's syndrome or ischemic stroke, or associated with intracranial aneurysms. As intracranial aneurysms may rupture and lead to subarachnoid haemorrhage, the American Heart Association recommends performing magnetic resonance angiography (MRA) of intracranial arteries in patients with cervical artery FMD.

      Mesenteric and iliac arteries were examined during renal artery angiography and cervical arteries were systematically examined using ultrasonography. In the European Georges-Pompidou Hospital (HEGP) cohort (unpublished results), cervical arteries were not systematically examined. The prevalence of diagnosed multi-site FMD was 28.0% in the Zurich University Hospital study and 16.4% in HEGP patients. This is probably a bottom estimate because most cervical artery FMD lesions affect the C1-C2 segment of the carotid arteries, a segment difficult to examine using ultrasonography. In order to estimate study power and the number of patients needed, the prevalence is considered of multi-site FMD at 20-25%.
   3. Diagnosis

      The presence of renal artery FMD can be documented by the following non-invasive tests, in increasing order of accuracy: Doppler ultrasound, gadolinium-enhanced MRA, and computed tomographic angiography (CTA). Vasbinder et al. (2004) prospective multicenter comparative study found that CTA and MRA had reasonably good specificities for detecting renal artery stenosis due to FMD (92 and 84%, respectively). There is no published comparative study of non-invasive tests for detecting cervical artery FMD, although Doppler ultrasound may disclose irregular patterns of stenosis that are suggestive. CTA and MRA are probably more effective than ultrasonography for detecting lesions of the middle and distal portions of the carotid and vertebral arteries and may also document or rule out associated intracranial aneurysms.

      The commonly accepted gold standard for diagnosing renal artery FMD is intra-arterial angiogram with digital subtraction. However, this invasive test should be reserved for patients in whom it is clinically justified to proceed with revascularization in the same procedure. Stenosis quantification is, however, frequently difficult in medial FMD with the "string-of-beads" appearance because multiple web-like defects are often present in patients with FMD, contributing to clinically significant stenoses that may not be apparent on angiography.
   4. Management

      The value of treatment has not been established for renal artery FMD without hypertension. The management of hypertension associated with renal artery FMD involves revascularization and/or antihypertensive medication. Current recommendations reflect the knowledge acquired concerning atherosclerotic renovascular hypertension, although indications for balloon angioplasty are wider in FMD than in atherosclerotic renovascular disease because the BP outcome of angioplasty is more favourable in FMD than in atherosclerosis. Revascularization is recommended for patients with hemodynamically significant renal artery stenosis - i.e. with bilateral stenoses or a unilateral stenosis causing more than 60% reduction in luminal diameter - and accelerated hypertension, resistant hypertension, malignant hypertension, hypertension with an unexplained unilateral small kidney, and hypertension with intolerance to medication. It is also useful in young patients with recent-onset hypertension and hemodynamically significant renal artery stenosis due to FMD: in these cases the goal is to cure hypertension. The standard revascularization procedure is balloon angioplasty with bailout stent placement if necessary. Surgical reconstruction is indicated for patients with complex FMD that extends to segmental arteries and those with macroaneurysms. Antihypertensive drug treatment is indicated for patients with long-standing hypertension or in those with persistent hypertension following revascularization.

      Data on management of patients with symptomatic carotid or vertebral artery FMD are scarce. Carotid or vertebral artery dissections are usually treated with anticoagulation. In very rare patients with expanding or symptomatic pseudo-aneurysm, percutaneous angioplasty or surgical repair can be considered.
   5. Progression in FMD

      Renal artery FMD may progress to more severe stenosis and to renal atrophy, and/or to stenoses affecting more arteries within or outside the renal vasculature. The risk of progression as assessed from available studies was probably overestimated because documentation of progression was obtained from angiography, a procedure which is not routinely undertaken in patients with favourable clinical and biological outcomes. The disease is progressive, however, and a Slovut and Olin overview (2004) stated that patients with FMD should undergo yearly duplex ultrasonography to detect progression of disease, restenosis, or loss of kidney volume.

      There are very few data on prognosis of patients with symptomatic carotid or vertebral artery FMD. The risk of arterial disease progression over time is unknown. The risk of ischemic stroke ranged from 0 to about 3% per year in the few studies which assessed that issue.
   6. Best Clinical Practice

      Published recommendations include:
      * Screening for any cause of secondary hypertension - including renal artery FMD - in case of juvenile, grade 3, malignant or resistant hypertension
      * Irrespective of the severity of hypertension, screening for renal artery stenosis in cases with a clinical clue for the condition, such as the presence of paraombilical bruit or of asymmetrical kidneys
      * Screening for cervical and intracranial FMD in case of renal artery FMD
      * Renal revascularization in case of hemodynamic stenosis associated with hypertension in a patient aged 30 or less, or associated with accelerated, malignant or resistant hypertension, or associated with a small kidney or treatment intolerance
      * In case of documented renal artery FMD, providing follow-up of blood pressure (BP), renal function and kidney height using ultrasonography on a yearly basis or in case of hypertension persistence or recurrence following revascularization, or in case with a poor control of BP.

      In case of renal artery FMD progression, further renal imaging tests and renal revascularization may be considered in accordance with the above indications for revascularization. The investigators also consider that documented progression of renal artery FMD is an indication to screen for new lesions or progression of pre-existing lesions in cervical arteries.
   7. Genetic factors

      FMD appears to be a familial disease in 10% of cases (OMIM #135580). The occurrence of renal FMD in sib pairs or identical twins first suggested its possible inheritability. Our retrospective analysis of 104 patients with renal FMD showed a prevalence of 11% for familial cases, i.e. 11% of cases had at least one sibling with angiographic evidence of renal artery FMD. Using high-resolution echo-tracking, elevated echo-tracking scores of the carotid artery in first-degree relatives of index cases are also found. FMD is diagnosed earlier, renal artery lesions are more frequently bilateral, and FMD lesions are more frequently found in extra-renal arteries in familial than in apparently sporadic cases. The presence of an underlying genetic disease could therefore be associated with disease progression in FMD.

      The investigators have already collected lymphocyte DNA and assessed baseline characteristics, including renal artery morphology, in about 400 patients with renal artery FMD who gave informed written consent to a familial study of renal artery FMD (Sponsor INSERM, RBM#00-028, CPP Paris-Cochin). Data from patients included in this previous study will be used for an extended case-control study.
   8. Justification for an extended genome-wide study

   As indicated above, several arguments exist for the presence of susceptibility genes for FMD. Despite this evidence, only limited and negative candidate gene studies have been conducted up to now, probably because of the low frequency of the disease, its phenotypic heterogeneity and the absence of large national or international collection of affected subjects. In the meantime, the knowledge acquired on the structure and variations of the human genes by the Human Genome Project and the possibility of rapidly genotyping hundreds or thousands of single nucleotide polymorphisms (SNPs) through high-throughput technologies facilitate large case-control studies. Case control studies are indeed powerful methods to investigate the implication of genetic SNPs in complex traits. It can be applied either to candidate genes or through the microarray technology. With this technique, it can test three to five hundreds of thousands SNPs (300 to 500K) along the human genome (genome-wide association (GWA) studies). Compared to candidate genes, GW-SNPs typing offers the advantage that new pathways can be uncovered. Whereas this strategy usually requires large number of cases and controls in complex traits, it has also been used with success for some categorical traits in experimental settings investigating a small number of well characterized subjects. To our knowledge, GWA studies have never been performed for FMD. The collection of 400 FMD at HEGP together with the national prospective study now makes this objective realistic.
2. Objectives of the ARCADIA registry

   1. To collect standardized clinical, radiological, and biological data in patients with FMD through a national registry.

      The prospective collection of clinical, radiological and biological standardized records should lead in a short period of time to a unique source of well-phenotyped FMD cases that could help to standardize diagnostic and therapeutic procedures at the national level. This unique database and collaboration between centres will greatly stimulate basic, clinical and therapeutic research and will help in the identification of new pathophysiological mechanisms.

      This collection of symptomatic patients will be established from centres dedicated to hypertension care (renovascular lesions) or to cerebrovascular diseases care (cervical lesions). It is expected to recruit 400 patients presenting with renovascular lesions and 100 patients presenting with cervical FMD over three years.
   2. To estimate the prevalence of multiple sites disease, i.e. the prevalence of cervical artery FMD in patients with renal artery FMD and vice versa.

      As indicated above, screening for cervicocranial FMD is currently recommended in patients with renal FMD. Although there is no similar recommendation to screen for renal artery FMD in patients with cervical FMD, such screening is required at least in patients with high blood pressure, i.e. with a clue for renovascular disease. It is also useful in cases without definite hypertension as the presence of renal artery FMD lesions would also help to confirm the FMD nature of cervical lesions. The investigators therefore consider that a non-invasive investigation of renal arteries in patients with probable or suspected cervical FMD reasonably falls within best clinical practices.
   3. To identify susceptibility genes for renal artery FMD and polymorphisms that could play a role in disease progression and to assess potential phenotype-genotype correlations.
   4. To organize a clinical, radiological and biological database and a biobank that will constitute a unique resource to initiate further clinical research.

Our goal is to share a common anonymous standardized database, the items of which have been accepted by the participating centres, that will serve as a unique national FMD database available for all Hypertension Reference Centres (ESH Hypertension Reference Centres) and vascular neurologists involved in the study. The creation and the development of this database will be a unique tool for future national studies and will stimulate similar initiatives at the European level.

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal or craniocervical fibromuscular dysplasia diagnosed during the 4 years before inclusion
* Who understood and signed inform consent form
* Affiliated to the French health insurance system
* The fibromuscular dysplasia is documented by imaging (angiography, CT-angiography, MR-angiography) of less than 4 years and validated by a radiologist investigator

Exclusion Criteria:

* Patient with renal or craniocervical atherosclerosis, or inflammatory vascular disease as dominant pathological features
* Patient with renal or craniocervical arteries dissection or aneurysm without any other evidence of fibromuscular dysplasia
* Patient under 18 or under tutorship
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal or craniocervical fibromuscular dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2009-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of multisite fibromuscular dysplasia confirmed by imaging | Inclusion
  FMD lesions discovered outside the symptomatic site

SECONDARY OUTCOMES:
Clinical characteristics associated with multisite fibromuscular dysplasia | Inclusion
Single nucleotide polymorphisms | Inclusion
  Assessed by genome-wide association

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Francois Plouin, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (17):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium
- France (16):
  - CHU de Bordeaux hopital Saint-Andre, Bordeaux, Aquitaine-Limousin-Poitou-Charentes
  - CHU de Clermont-Ferrand hopital Gabriel-Montpied, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU de Grenoble hopital Albert-Michallon, La Tronche, Auvergne-Rhône-Alpes
  - CHU de Nancy institut Louis-Mathieu, Vandœuvre-lès-Nancy, Grand Est
  - CHRU de Lille hopital cardiologique, Lille, Hauts-de-France
  - CHRU de Lille hopital Roger-Salengro, Lille, Hauts-de-France
  - CHU de Caen hopital Cote de Nacre, Caen, Normandy
  - CHU de Toulouse hopital Rangueil, Toulouse, Occitanie
  - AP-HM hopital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de Versailles hopital Andre Mignot, Le Chesnay, Île-de-France Region
  - AP-HP hopital Lariboisiere, Paris, Île-de-France Region
  - AP-HP hopital Pitie-Salpetriere, Paris, Île-de-France Region
  - Centre hospitalier Sainte-Anne, Paris, Île-de-France Region
  - AP-HP hopital Bichat-Claude-Bernard, Paris, Île-de-France Region
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region
  - AP-HP hopital Tenon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Controlled access

REFERENCES:
- [Derived] Arnaud C, Boulanger M, Lorthioir A, Amar L, Azarine A, Boyer L, Chatellier G, Di Monaco S, Jeunemaitre X, Kastler A, Mousseaux E, Oppenheim C, Thony F, Persu A, Olin JW, Azizi M, Touze E; ARCADIA Co-investigators dagger. Male Sex Is Associated With Cervical Artery Dissection in Patients With Fibromuscular Dysplasia. J Am Heart Assoc. 2021 Jun;10(11):e018311. doi: 10.1161/JAHA.120.018311. Epub 2021 May 17. PMID 33998257
- [Derived] Plouin PF, Baguet JP, Thony F, Ormezzano O, Azarine A, Silhol F, Oppenheim C, Bouhanick B, Boyer L, Persu A, Hammer F, Gosse P, Mounier-Vehier C, Le Hello C, Jeunemaitre X, Azizi M, Amar L, Chatellier G, Mousseaux E, Touze E; ARCADIA Investigators. High Prevalence of Multiple Arterial Bed Lesions in Patients With Fibromuscular Dysplasia: The ARCADIA Registry (Assessment of Renal and Cervical Artery Dysplasia). Hypertension. 2017 Sep;70(3):652-658. doi: 10.1161/HYPERTENSIONAHA.117.09539. Epub 2017 Jul 17. PMID 28716989